CLINICAL TRIAL: NCT00187590
Title: A Case Management Intervention to Prevent ER Visits in HIV-infected Persons
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention was taken up as a standard of care.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMC200517
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: HIV
Keywords: HIV; case management

ARMS (2):
- Intervention (Experimental): Phone call after an ER visit.
  Interventions: Behavioral: Case manager phone call after an ER visit
- Control (No Intervention): No phone call after an ER visit.

INTERVENTIONS:
Behavioral: Case manager phone call after an ER visit
  Arms: Intervention

SUMMARY:
Case management has become an integral part of HIV care. There is little science however demonstrating its effectiveness. This is a randomized, controlled trial of a phone call intervention after an ER visit to see if this can reduce further ER visits, hospitalizations, deaths, and cost.

DETAILED DESCRIPTION:
One year retrospective look at outcome measures followed by a one year trial of a phone call after each ER visit in half of the group. Outcomes measured are cost, ER visits, hospitalizations, death, length of stay. Adults only, English or Spanish, questionnaire on depression, appointments, drug use with referral to case management services, drug rehab services, or followup appointments. Time for intervention is recorded to estimate cost.

ELIGIBILITY:
Inclusion Criteria:

* Patient in our clinic as of 4-1-04

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2004-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Death, hospitalizations, ER visits, LOS | 1 year

SECONDARY OUTCOMES:
Cost | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roger B Mortimer, MD, Principal Investigator — UCSF-Fresno Medical Eduction Program
Locations (1):
- University Medical Center, Fresno, California, United States